CLINICAL TRIAL: NCT04961931
Title: Effect of Empagliflozin on Urinary Excretion of Adenosine and on Markers of Osteocyte Function and Glomerular Damage in Diabetic and Non-diabetic Patients With Chronic Kidney Disease
Brief Title: Effect of Empagliflozin on Urinary Excretion of Adenosine and Osteocyte Function in Patients With Chronic Kidney Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Michal Nowicki, Professor, Medical University of Lodz
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EMPA - 1 - AMZ
Record Dates: First submitted 2021-06-30; First posted 2021-07-14 (Actual); Last update posted 2021-07-14 (Actual); Status verified 2021-07

CONDITIONS: Chronic Kidney Disease stage3
Keywords: SGLT2 inhibitors; adenosine; calcium-phosphate metabolism; chronic kidney disease; diabetes; non-diabetes; albuminuria
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Albuminuria | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: The study will be prospective, interventional and will be conducted in two parallel groups selected on the basis of clinical diagnosis (diabetic nephropathy or other chronic nephropathies).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- diabetes group (Other): After qualifying for the study subjects with diabetes and chornic kidney disease received oral empagliflozin 10 mg once daily for 7 days.
  Interventions: Drug: Empagliflozin 10 MG
- non-diabetes group (Other): After qualifying for the study subjects with chronic kidney disease without diabetes received oral empagliflozin 10 mg once daily for 7 days.
  Interventions: Drug: Empagliflozin 10 MG
- control (Other): After qualifying for the study healthy subjects received oral empagliflozin 10 mg once daily for 7 days.
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — After qualifying for the study all subjects received oral empagliflozin 10 mg once daily for 7 days.
  Other Names: Jardiance

SUMMARY:
Sodium-glucose cotransporter 2 (SGLT2) inhibitors are the newest class of orally drugs for the treatment of type 2 diabetes. These drugs decrease plasma glucose levels by inhibiting its reabsorption in the proximal tubules of the kidney. They have an attractive clinical efficacy profile, including glycemic control, weight loss, and lowering blood pressure. SGLT2 inhibitors have also been reported to reduce the risk of severe adverse cardiovascular events and progression of diabetic kidney disease. SGLT2 is expressed in the kidney, while its expression in other tissues is most likely negligible or absent.

SGLT2 dilates the supply vessels to the glomerulus thereby promoting hyperfiltration. In animal models SGLT2 has been shown to reduce the excretion of macular dense adenosine, which may contribute to the excessive glomerular filtration rate as a result of vasodilation of the afferent vessels. Adenosine, unlike other vascular regions, increases the tension in the walls of the vessels supplying blood to the glomerulus. The role of adenosine in humans in this regard is poorly defined, although treatment with empagliflozin has recently been shown to increase the urinary excretion of adenosine in type 1 diabetic patients with controlled hyperglycemia. Our working hypothesis is that the SGLT2 inhibitor empagliflozin may reduce the hyperfiltration of residual nephrons by increasing adenosine production, which affects the contraction of the afferent arterioles, and this effect occurs in various types of nephropathy.

In addition, it has been described that SGLT2 inhibitors may affect individual parameters of calcium-phosphate metabolism, leading to changes in bone mineral density and an increase in bone resorption marker SGLT2 inhibitors also stimulate renal, proximal phosphate reabsorption. Increased phosphate reabsorption triggers the secretion of fibroblast growth factor 23 (FGF23). FGF23 inhibits the production of 1,25-dihydroxyvitamin D (the biologically active form of vitamin D), which reduces the absorption of calcium from the gastrointestinal tract, thereby stimulating the secretion of parathyroid hormone (PTH). In the conducted studies, it was found that SGLT2 inhibitors increase the concentration of serum phosphorus, FGF23 in the plasma and PTH in the plasma, while lowering the level of 1,25-dihydroxyvitamin D.

DETAILED DESCRIPTION:
The study will be prospective, interventional and will be conducted in two parallel groups selected on the basis of clinical diagnosis. It is planned to enroll 60 patients aged 18-70 years under outpatient nephrological care, with impaired excretory function of the kidneys (eGFR 20-60 ml / min / 1.73 m3), with proteinuria above 0.5-3 g / l in the morning urine sample , including 30 nondiabetic and 30 diabetic patients t.2 and 20 healthy control subjects (no microalbuminuria and no impaired renal function with eGFR> 90 ml / min / 1.73m3). After the patients are familiarized with the objectives of the study and the informed consent signed, the following procedures will be performed.

After signing the consent, basic biochemical tests will be performed in both groups to assess the concentration of protein, albumin, calcium, phosphate, adenosine and creatinine in the morning urine sample, creatinine, calcium, phosphate, PTH, bacterial alkaline phosphatase (BAP), 1.25 vitamin D, sclerostins, FGF23, serum Klotho proteins, eGFR, plasma glucose. The tests will be repeated after 7 days of taking empagliflozin in a dose of 10 mg a day. On days 1 and 7, patients will be given an intravenous glucose 5% solution at a dose of 240 mg glucose / kg body weight in the first 15 minutes to induce a controlled hyperglycaemia state in the first 15 minutes, this will increase their blood glucose by 125 mg / dL in 15 minutes followed by 10-12 mg glucose / kg body weight, under glycemic control to maintain a concentration of 200 mg / dL ± 5% for 120 minutes. Stability of serum glucose levels during this period will be maintained by adjusting the rate of intravenous glucose infusion based on blood glucose measurements, every 15 minutes. After 2 hours of infusion, additional blood will be drawn for the determination of glucose and renal parameters and after 100 ml of urine for determination. adenosine, albumin and creatinine concentrations. In healthy subjects from the control group, the above basic blood and urine biochemical tests will be performed once.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes complicated by diabetic nephropathy (first group), non-diabetic nephropathy (second group) or healthy subjects
* Angiotensin-converting enzyme inhibitor or antagonists of angiotensin receptor blockers in the stable dose for the 4 months
* age 18 - 70 years
* stable clinical condition for the last 3 months
* GFR 25-60 ml / min / 1.73 m2
* proteinuria 0.5-3 g / day

Exclusion Criteria:

* diabetes mellitus other than t.2
* have taken SGLT2 inhibitors in the last 4 weeks or have ever had an intolerance to SGLT2 inhibitors in the past
* acute kidney damage
* systolic blood pressure <90 mmHg
* Cancer
* acute inflammation
* liver failure
* heart failure> 2. NYHA grade
* pregnancy
* patients with impaired consciousness and testers with insufficient management in the past.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
albuminuria | 7 days
  ratio of albumin to creatinine in urine in mg/g
serum calcium concentration | 7 days
  serum calcium level in mmol/l
urine calcium concentration | 7 days
  level of calcium in urine in mmol/l
urine adenosine | 7 days
  adenosine in urine in µmol/mmol creatinine
urine phosphorus concetration | 7 days
  serum phosphorus level in mmol/l
serum Fibroblast growth factor 23 concentration | 7 days
  serum Fibroblast growth factor 23 level in pg/ml
serum parathormone concentration | 7 days
  serum parathormone level in pg/ml
serum Klotho concentration | 7 days
  serum Klotho level in ng/ml
serum Bone alkaline phosphatase concentration | 7 days
  serum Bone alkaline phosphatase level in µg/l
serum 1,25(OH)2D concentration | 7 days
  serum 1,25(OH)2D level in pg/ml
serum sclerostin concentration | 7 days
  serum sclerostin level in pmol/l
urine phosphorus concetration | 7 days
  phosphorus in urine in mmol/l

CONTACTS AND LOCATIONS:
Overall Officials: Ireneusz Staroń, Study Chair — Medical University of Lodz
Locations (1):
- Department of Nephrology, Hypertension and Kidney Transplantation, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No